CLINICAL TRIAL: NCT06136702
Title: EarLy dEtection of cerVical cAncer in Hard-to-reach Populations of Women Through Portable and Point-of-care HPV TEsting Acceptability Study
Brief Title: ELEVATE Acceptability Study
Acronym: ELEVATE AS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Collaborators: Horizon 2020 - European Commission (Other); Universidade Nova de Lisboa (Other); Universidad de Cuenca (Other); Hospital de Cancer de Barretos - Fundacao Pio XII (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ONZ-2022-0326
Record Dates: First submitted 2023-10-20; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cervical Cancer; HPV Infection; Acceptability of Health Care
Keywords: cervical cancer; screening; self-sampling; HPV; acceptability; hard-to-reach; underscreened; community-based
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Longitudinal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational session and follow-up assessment (Active Comparator): A community-based researcher will educate women about sexual health and cervical cancer by using the materials that will be developed by the ELEVATE team. Women will be informed about cervical cancer screening (pap smear) and about where they can obtain these services off-site (health facilities). Furthermore, a self-administrated questionnaire is applied to assess current knowledge, willingness to get screened (clinically collected sample) and uptake
  Interventions: Behavioral: Educational session; Behavioral: Follow-up assessment
- Educational session, self-sampling and follow-up assessment (Experimental): A community-based researcher will educate women about sexual health and cervical cancer by using the materials that will be developed by the ELEVATE team. In addition, women will receive information about self-sampling and will be instructed by the community-based researcher on how to take a self-sample using an illustrative cartoon. Women will then be invited to take a sample on-site. The researcher will collect all samples for analysis by an HPV test in a lab. Sample analysis is expected to take 2 weeks time.
  Interventions: Behavioral: Educational session; Behavioral: Self-sampling; Behavioral: Follow-up assessment

INTERVENTIONS:
Behavioral: Educational session — A community-based researcher will educate women about sexual health and cervical cancer by using the materials that will be developed by the ELEVATE team. Women will be informed about cervical cancer screening (pap smear) and about where they can obtain these services off-site (health facilities). Furthermore, a self-administrated questionnaire is applied to assess current knowledge, willingness to get screened (clinically collected sample) and uptake.
Behavioral: Self-sampling — Women will receive information about self-sampling and will be instructed by the community-based researcher on how to take a self-sample using an illustrative cartoon. Women will then be invited to take a sample on-site, to measure the uptake of the self-sampling test (% of women who take the self-sample). Furthermore, two self-administrated questionnaires are applied to 1) assess attitudes regarding self-sampling (pre-intervention), and 2) assess users' experience regarding self-sampling (post-intervention). The researcher will collect all samples for analysis by an HPV test in a lab. Sample analysis is expected to take 2 weeks time. All women will be contacted 1-2 weeks after the self-sample taking to inform them on their test result.
  Arms: Educational session, self-sampling and follow-up assessment
Behavioral: Follow-up assessment — To gauge the knowledge on cervical cancer screening after the educational session and to verify whether they got a pap smear, a 3-month follow-up is proposed for all women receiving an educational session (arm 1) and all women receiving an educational session and a self-sample (arm 2), because all women, whether or not invited for self-sampling, are provided information on where to get screened, although there is no formal referral to screening services.

SUMMARY:
This study includes a community-based, two-arm prospective acceptability study, whereby arm 1 consists of an educational session on sexual health and cervical cancer (screening) and a follow-up assessment after 3 months. Arm 2 consists of an educational session on sexual health and cervical cancer (screening) and self-sampling, additionally women will be asked to take a self-sample on-site, followed by a follow-up assessment after 3 months. Attitudes, uptake and users' experiences related to the use of a HPV self-sampling test will be assessed, additionally, the impact on looking for follow up care of self-sampling with standard cervical screening strategies will be assessed and finally the feasibility of an HPV self-sampling in hard-to-reach groups versus educational sessions and standard care will be compared (arm 1 and 2).

DETAILED DESCRIPTION:
ELEVATE, a five-year project conducted by an international research alliance led by Ghent University, aims to develop a new test and approach for cervical cancer screening in hard-to-reach populations. The test will combine self-sampling with a new low-cost, portable measurement device and will be validated in dedicated screening trials in Belgium, Brazil, Ecuador, and Portugal. The ELEVATE project targets women in Europe and Latin America who have never been screened or are not regularly screened. These women have a higher risk of developing cervical cancer. The project is supported by the European Union's Horizon 2020 Framework Programme for Research and Innovation Action, project number 825747.

To address the gaps in cervical cancer screening, the ELEVATE project is developing a screening strategy to make cervical screening more accessible to hard-to-reach women. This strategy will include the introduction of a new on-site HPV self-sampling screening tool and a portable testing device, able to detect the presence of HPV and cancer biomarker proteins. This portable, low-cost, on-site HPV testing tool will allow to streamline follow-up care for women at risk of developing cervical cancer.

This study is part of the ELEVATE project and takes place in hard-to-reach communities, focusing on socio-economically vulnerable women to assess the acceptability of educational sessions and self-sampling in these communities. This study includes a two-arm prospective acceptability study, whereby arm 1 consists of an educational session on sexual health and cervical cancer (screening) and a follow-up assessment after 3 months. Arm 2 consists of an educational session on sexual health and cervical cancer (screening) and self-sampling, additionally women will be asked to take a self-sample on-site, followed by a follow-up assessment after 3 months. Attitudes, uptake and users' experiences related to the use of a HPV self-sampling test will be assessed, additionally, the impact on looking for follow up care of self-sampling with standard cervical screening strategies will be assessed and finally the feasibility of an HPV self-sampling in hard-to-reach groups versus educational sessions and standard care will be compared (arm 1 and 2).

ELIGIBILITY:
Inclusion Criteria:

* are between the ages of 25 to 65 years of age, in line with the European Guidelines for initiating and stopping cervical cancer screening
* (ever been) sexually active;
* not diagnosed or in treatment for cervical cancer;
* not having had a hysterectomy
* not being pregnant
* Speaking the local language

Exclusion Criteria:

* younger than 25 years old or older than 65 years old
* diagnosed or in treatment for cervical cancer
* having had a hysterectomy
* being pregnant

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1048 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Uptake of cervical cancer screening | First encounter (day 0) and 3 months follow-up (day 90)
  Compare the on-site uptake of self-sampling (arm2) with uptake of standard care (follow-up of arm1)

SECONDARY OUTCOMES:
Attitudes towards HPV self-sampling | First encounter (day 0)
  Attitudes towards self-sampling: reasons to accept/decline the self-sample; advantages and disadvantages versus conventional screening.
User's experiences of HPV self-sampling | First encounter (day 0)
  User experiences among those who took a self-sample (easy/difficult; painless/painfull; trustworthy/untrusty; etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Vega Crespo, Principal Investigator — Universidad de Cuenca; Adhemar Longatto, Principal Investigator — Barretos Cancer Hospital; Sónia Dias, Principal Investigator — Universidade Nova de Lisboa; Olivier Degomme, Principal Investigator — University Ghent
Locations (4):
- International centre for reproductive health, Ghent, East-Flanders, Belgium
- Barretos Cancer Hospital - Fundação Pio XII, Barretos, Brazil
- Universidad de Cuenca, Cuenca, Ecuador
- Escola Nacional de Saúde Pública da Universidade NOVA de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

DOCUMENTS (2):
  • Study Protocol (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT06136702/Prot_000.pdf
  • Informed Consent Form (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT06136702/ICF_001.pdf